CLINICAL TRIAL: NCT01429558
Title: Electrophysiological Recording for Patients Receiving Deep Brain Stimulation Electrode for Treatment-resistant Obsessive-compulsive Disorder
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Jean-Philippe Langevin, Assistant clinical professor of surgery, University of Arizona
Other Study IDs: 11-0290-03
Record Dates: First submitted 2011-09-04; First posted 2011-09-07 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Obsessive-compulsive Disorder
Keywords: treatment resistant obsessive-compulsive disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this project is to study live recordings from neuronal population of the human nucleus accumbens during the implantation of deep brain stimulation (DBS) electrodes for the treatment-resistant obsessive compulsive disorder (OCD). The central aim of this project is to determine if intra-operative electrophysiological data can confirm that the electrode is located in the nucleus accumbens. This confirmation could allow the placement of the DBS electrodes with a higher degree of precision. An additional aim of this project will be to study the activity of the neuronal population of the nucleus accumbens while a subject is presented with a task involving an unexpected reward.

The investigators central hypothesis is that unexpected reward will be associated with increase firing and synchrony in the neuronal population. This will translate into recordable increase activity in the investigators region of interest and therefore confirm the proper placement of the electrode.

This study enrolled 2 subjects, with 1 subject completing the protocol showing the feasibility of the experiment. There were electrophysiological variations with the task presented but no conclusion could be drawn given the small sample size.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-resistant OCD
* Failure of psychotherapy
* Failure of pharmacotherapy
* Meets inclusion criteria for DBS implant in OCD

Exclusion Criteria:

* Significant substance use disorder
* Significant personality disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects in this study are suffering from treatment-resistant OCD
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States